CLINICAL TRIAL: NCT05564520
Title: Etude Multicentrique Internationale Sur le déficit en Lipin-1
Brief Title: International Multicenter Study on Lipin-1 Deficiency
Acronym: LIPIN1
Status: Recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HJ-23-LIPIN1
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Lipin-1 Deficiency
Keywords: Inherited Metabolic Diseases; enzymatic deficiency; rhabdomyolysis
MeSH Terms: conditions — Rhabdomyolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
LIPIN1 is an international registry that allows the collection of data on the follow-up, management and treatment of patients with Lipin-1 deficiency.

DETAILED DESCRIPTION:
This study evaluates survival, cardiac function, quality of life, fatigability, treatment tolerance and comparison of the efficacy of different current treatments in patients with Lipin-1 deficiency.

ELIGIBILITY:
Inclusion Criteria:

Patient at least 12 months with Lipin1 deficiency confirmed by molecular biology (two causal mutations in the LPIN1 gene)

Exclusion Criteria:

Opposition of the patient or his parents to participate to the study

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with lipin1 deficit with two mutations on the LIPIN1 gene and having undergone acute rhabdomyolysis, 50 to 150 patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of survival in patients with Lipin-1 deficiency | According to routine care
  Patient survival as assessed by long-term follow-up

SECONDARY OUTCOMES:
Evaluation of cardiac function in patients with Lipin-1 deficiency | According to routine care
  Cardiac function, assessed by cardiographic ultrasound
Comparison of the effectiveness of different current treatments in patients with Lipin-1 deficiency | According to routine care
  Comparison of the number of severe rhabdomyolysis and biological assessment (CPK measurement performed as part of care) in patients
Evaluation of the quality of life of patients with Lipin-1 deficiency | According to routine care
  Quality of life, assessed by standardized questionnaires
Evaluation of the tolerance of treatments in patients with Lipin-1 deficiency. | According to routine care
  Treatment side effects, assessed by abdominal pain, skin allergy and other adverse effects
Evaluation the fatigability of patients with Lipin-1 deficiency | According to routine care
  Exercise capacity, assessed by walking tests

CONTACTS AND LOCATIONS:
Overall Officials: Pascale De Lonlay, Pr, Principal Investigator — Necker Hospital; Hortense De Calbiac, Ph.D., Study Chair — Institut Imagine; Caroline Tuchmann-Durand, Pharm D, Study Chair — Institut Imagine
Locations (1):
- Necker - Enfants Malades Hospital, Paris, France